CLINICAL TRIAL: NCT07162857
Title: The Value of Critical Care Ultrasound and Noninvasive Cardiac Output Monitoring in Guiding Fluid Resuscitation for Septic Shock in the Emergency Department
Brief Title: Guiding Fluid Resuscitation in Septic Shock: Ultrasound vs. Noninvasive Cardiac Output Monitoring
Acronym: CUS-NICOM-SS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mai Xiaowei (Other)
Collaborators: Guangzhou Panyu Central Hospital (Other)
Responsible Party: Sponsor-Investigator, Mai Xiaowei, Emergency Department Attending Physician，Guangzhou Panyu Central Hospital, Guangzhou Panyu Central Hospital
Organization: Guangzhou Panyu Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PYRC-2023-088; 2024-Z04-020 (Other Grant/Funding Number: Guangzhou Panyu District Science and Technology Program Project); PYRC-2023-088 (Other: Medical Ethics Committee of Panyu Central Hospital)
Record Dates: First submitted 2025-08-16; First posted 2025-09-09 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Septic Shock
Keywords: critical care ultrasound; noninvasive cardiac output monitoring; eptic shock; fluid resuscitation
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Critical Care Ultrasound Group (Experimental): patients underwent immediate bedside assessment using a Philips EPIQ 5 color Doppler ultrasound system equipped with both phased-array (1.5-4.0 MHz) and convex-array (2.0-5.0 MHz) transducers. The initial ultrasound evaluation was completed within 10 minutes of enrollment and included comprehensive hemodynamic monitoring: inferior vena cava diameter (IVC) and collapsibility index (IVC-CI) for volume status assessment, left ventricular ejection fraction (LVEF) and end-diastolic volume (LVEDV) for cardiac function evaluation, ventricular wall motion analysis, along with pulmonary B-line quantification to assess pulmonary edema.
  Interventions: Device: Ultrasonic technology
- Non-Invasive Cardiac Output Monitoring (NICOM) Group (Experimental): In the noninvasive cardiac output monitoring group, continuous hemodynamic assessment was performed using the NICOM system based on thoracic bioreactance technology.
  Interventions: Device: non-invasive cardiac output monitoring

INTERVENTIONS:
Device: non-invasive cardiac output monitoring — Monitoring commenced immediately after enrollment, with baseline parameters recorded after signal stabilization (≤5 minutes), including cardiac output (CO), stroke volume (SV), stroke volume variation (SVV), and systemic vascular resistance (SVR). The system automatically updated these parameters every 30 seconds and displayed them in real-time on the monitor screen. Fluid resuscitation was dynamically adjusted according to these continuous measurements until achieving the predefined therapeutic targets.
  Arms: Non-Invasive Cardiac Output Monitoring (NICOM) Group
Device: Ultrasonic technology — In the critical care ultrasound group, patients underwent immediate bedside This protocol ensured real-time, comprehensive evaluation of both cardiac function and fluid status to guide resuscitation.Ultrasound reassessment was performed every 1-2 hours to dynamically adjust both the volume and rate of fluid administration until predefined resuscitation targets were achieved.
  Arms: Critical Care Ultrasound Group

SUMMARY:
This randomized controlled study investigates the value of critical care ultrasound and non-invasive cardiac output monitoring in guiding fluid resuscitation for patients with septic shock in the emergency department. A total of 60 patients are randomly assigned to receive either ultrasound-guided or NICOM-guided fluid management, with both groups receiving standard sepsis care according to the 2021 Surviving Sepsis Campaign guidelines.

The study aims to evaluate whether these monitoring modalities can optimize hemodynamic management, improve prognosis, and support clinical decision-making in emergency settings. Primary and secondary outcomes include early resuscitation efficacy (time to achieve mean arterial pressure ≥65 mmHg and lactate clearance), total fluid volume within the first 6 hours, incidence of complications (pulmonary edema, renal injury, ARDS), length of stay in the emergency department and hospital, and 28-day mortality.

By comparing these two approaches, this study seeks to provide evidence for selecting appropriate monitoring tools to achieve precise and individualized fluid resuscitation in septic shock.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled trial conducted in the Emergency Department of Guangzhou Panyu Central Hospital. Eligible adult patients with septic shock, admitted between july 2023 and july 2025, were enrolled after informed consent. Demographic and baseline clinical data, including age, gender, comorbidities, mean arterial pressure, baseline lactate, and vital signs, were collected at enrollment.

A total of 60 patients were randomly assigned to one of two intervention groups using block randomization generated by SPSS software, with allocation concealed by sealed envelopes.

* Critical Care Ultrasound Group: Patients underwent bedside ultrasound assessment, including inferior vena cava diameter and collapsibility index (IVC-CI), left ventricular ejection fraction (LVEF), left ventricular end-diastolic volume (LVEDV), ventricular wall motion, and pulmonary B-lines, to guide individualized fluid resuscitation. Ultrasound evaluations were repeated every 1-2 hours until resuscitation targets were achieved.
* Non-Invasive Cardiac Output Monitoring (NICOM) Group: Patients received continuous hemodynamic monitoring using thoracic bioreactance technology. Parameters including cardiac output (CO), stroke volume (SV), stroke volume variation (SVV), and systemic vascular resistance (SVR) were continuously recorded and used to guide fluid therapy adjustments until resuscitation targets were achieved.

In both groups, all patients received standard septic shock management based on the 2021 Surviving Sepsis Campaign guidelines, including early antibiotics, vasopressor therapy, and organ support. Outcomes recorded included total fluid volume within the first 6 hours, time to resuscitation targets, complications (e.g., pulmonary edema, renal injury, ARDS), emergency department and hospital length of stay, 28-day mortality, and adverse events (e.g., arrhythmias, anaphylaxis).

ELIGIBILITY:
Inclusion criteria:

1. diagnosis of septic shock in accordance with the Surviving Sepsis Campaign International ;
2. receipt of initial fluid resuscitation in the emergency department with a hospital stay of at least 6 hours;
3. age ≥ 18 years;
4. provision of informed consent.

Excluded criteria:

1. contraindications to rapid fluid administration (e.g., end-stage renal disease, end-stage heart failure, acute pulmonary edema);
2. inability to comply with treatment, such as patients with severe trauma, burns, cancer undergoing chemotherapy, pregnant or lactating women, and those with mental illness;
3. withdrawal from treatment or transfer to another facility within 24 hours of admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-07-05 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
28-day mortality rate | 28 days from enrollment
  Proportion of patients who die within 28 days after enrollment. Mortality will be assessed using hospital records and survival follow-up.
28-Day Survival | 28 days from enrollment
  Proportion of patients who survive at 28 days after enrollment.

SECONDARY OUTCOMES:
ICU hospitalization time | From enrollment to the end of treatment at 4 weeks
  Number of days each patient remains in the intensive care unit (ICU) during the study period.
Use of Mechanical Ventilation | From enrollment to the end of treatment at 4 weeks
  Proportion of patients requiring invasive mechanical ventilation during hospitalization.
Duration of Mechanical Ventilation | From enrollment to the end of treatment at 4 weeks
  Number of days of invasive mechanical ventilation among patients who required ventilatory support.
Use of Vasopressor Therapy | From enrollment to the end of treatment at 4 weeks
  Proportion of patients requiring vasopressor therapy (e.g., norepinephrine, dopamine).
Time to Achieve Mean Arterial Pressure ≥65 mmHg | Within the first 6 hours after enrollment
  Time in minutes required from enrollment to reach a mean arterial pressure ≥65 mmHg.
Incidence of Pulmonary Edema | Within 28 days after enrollment
  Proportion of patients who develop pulmonary edema during hospitalization.
Proportion of Patients With Lactate Reduction ≥20% From Baseline | Within the first 6 hours after enrollment
  Percentage of patients whose serum lactate level decreased by ≥20% compared with baseline.
Proportion of Patients With Lactate Clearance ≥10% | Within the first 6 hours after enrollment
  Percentage of patients achieving lactate clearance ≥10% from baseline.
Incidence of Acute Kidney Injury (AKI) | Within 28 days after enrollment
  Proportion of patients who develop acute kidney injury, defined according to KDIGO criteria.
Incidence of Acute Respiratory Distress Syndrome (ARDS) | Within 28 days after enrollment
  Proportion of patients who develop ARDS during hospitalization, defined according to the Berlin definition.

CONTACTS AND LOCATIONS:
Overall Officials: yingshen wen, Principal Investigator — Guangzhou Panyu Central Hospital, Guangzhou, Guangdong , China
Locations (1):
- Panyu Central Hospital Affiliated to Guangzhou Medical University, Guangzhou, Guangdong, China

DOCUMENTS (2):
  • Study Protocol (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT07162857/Prot_002.pdf
  • Informed Consent Form (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT07162857/ICF_001.pdf